CLINICAL TRIAL: NCT07085884
Title: A Comprehensive Intervention Program of Static-dynamic Balance Training Combined With Reminiscence Therapy on the Level of Healthy Aging Among Older Adults in a Rural Community
Brief Title: Static-dynamic Balance Training Combined With Reminiscence Therapy
Acronym: SDBT-RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinyu Yang (Other)
Responsible Party: Sponsor-Investigator, Xinyu Yang, Master of Science, Huzhou University
Organization: Huzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-06-07
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Elderly (People Aged 65 or More); Rural Health
Keywords: Reminiscence therapy; balance training

STUDY DESIGN:
Intervention Model Description: The Theory of Planned Behavior (TPB), an extension of the Theory of Reasoned Action, evaluates individuals' intentions to engage in specific behaviors by considering both personal and social determinants of intention . TPB comprises four key constructs: attitude, subjective norm, perceived behavioral control, and behavioral intention. Previous studies have demonstrated that TPB has strong predictive validity for health behaviors requiring self-regulation, such as physical activity, making it a suitable framework for designing health interventions .
Who Masked: Participant, Outcomes Assessor
Masking Description: Data Analyst
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group received standardized health education and general exercise guidance delivered by trained staff at community centers. Biweekly, 40-minute, 12-week group sessions cover six topics: Static Balance Training Principles, Dynamic Equilibrium Skill Development, Psychosocial Adaptation Techniques, Fall Risk Mitigation Strategies, Home Environment Optimization, and Lifestyle Behavior Internalization, focusing on knowledge transmission and fundamental movement instruction.
- Intervention group (Experimental): The intervention lasted for 12 weeks. In odd-numbered weeks, a dual intervention model of "40-minute RT + 50-minute SDBT" was adopted to establish behavioral intentions, and behavioral attitudes and subjective norms were strengthened through RT.
  Interventions: Behavioral: The Static-Dynamic Balance Training Combined with Reminiscence Therapy

INTERVENTIONS:
Behavioral: The Static-Dynamic Balance Training Combined with Reminiscence Therapy — The intervention group received a 12-week SDBT-RT program, conducted twice weekly: 40-minute reminiscence therapy plus 50-minute balance training in odd weeks, and 50-minute balance training alone in even week.
  Arms: Intervention group

SUMMARY:
The SDBT-RT Program: A Holistic Approach for Rural Older Adults We developed the Static-Dynamic Balance Training Combined with Reminiscence Therapy (SDBT-RT) program to help older adults in rural communities adopt healthier habits. This program is rooted in the Theory of Planned Behavior , which emphasizes how attitudes, social norms, and perceived control influence behavior. It was designed specifically for rural contexts, considering local policies, lifestyle habits, social networks, and individual needs.

Key Components Expert Review & Pilot Testing Before launching, the program was refined by 5 experts in sports rehabilitation, medical psychology, geriatrics, health management, and nursing. A pilot study was conducted to ensure feasibility.

Static-Dynamic Balance Training (SDBT)

This physical training aims to improve stability and reduce fall risks. It includes:

10-Minute Warm-Up: Stretching wrists, hips, shoulders, knees, and ankles. 15-Minute Static Balance: Standing on both feet, tandem stance, and single-leg balance.

25-Minute Dynamic Balance: Walking normally, on narrow paths, and in tandem. Difficulty increases gradually with sensory challenges (e.g., distractions) and real-time guidance to build confidence .

Reminiscence Therapy (RT)

Based on Erikson's theory of psychosocial development , RT helps older adults reflect on life experiences to achieve psychological "integrity" (acceptance of life) over despair. Six structured themes guide discussions:

"Our Time," "My Happy Times," "Life Achievements," "Traditional Festivals," "My Hobbies," and "Nostalgic Memories." These activities foster optimism and self-acceptance, aligned with rural Chinese cultural practices .

Implementation Details Trained Staff: General practitioners, community health workers, and medical students underwent 1 month of training to lead sessions.

Group Structure: 32 participants were divided into 8-person groups and met at community centers (with multimedia facilities and green spaces) from 8:00-10:00 AM to align with their routines.

12-Week Intervention: Odd-Numbered Weeks: 40-minute RT + 50-minute SDBT. RT strengthens motivation (attitudes/norms), while SDBT improves physical control.

Even-Numbered Weeks: 50-minute SDBT only, focusing on skill mastery without cognitive overload.

Monitoring:

Observation Checklists and feedback forms tracked engagement and emotions. Implementation Fidelity Checklists ensured sessions followed protocols. Supervisors reviewed 20% of checklists weekly .

Behavior Log Forms recorded participants' health behaviors (e.g., supplement use, illnesses) to identify confounding factors.

Follow-Up: After the 12 weeks, participants received 4 weekly phone calls (5-10 minutes) to encourage home practice and address questions.

Safety & Adaptability Facilitators were trained to recognize fatigue or distress and adjust activities as needed.

Emergency protocols addressed physical/psychological incidents. Absent participants were contacted for makeup sessions, and adherence was prioritized.

This program integrates psychological reflection and physical training to empower rural older adults, fostering both mental well-being and functional independence. By tailoring interventions to local contexts and using evidence-based theories, SDBT-RT aims to create sustainable behavior change.

DETAILED DESCRIPTION:
The Static-Dynamic Balance Training Combined with Reminiscence Therapy (SDBT-RT) program, grounded in the Theory of Planned Behavior, was designed to promote positive health behaviors. Guided by TPB, an SDBT-RT program was developed, taking into account the rural community context-including local policies, lifestyle habits, and social networks-as well as individual-level characteristics. The formulation of a research protocol that incorporates the model's core constructs warrants further investigation. At the level of behavioral attitude, reminiscence therapy sessions are used to evoke positive memories, foster a constructive outlook on aging, and strengthen the belief that "participating in this program can enhance my well-being". At the subjective norm level, the group-based intervention delivered in community centers helps establish supportive social norms. Peer observation and interaction reduce perceived barriers to participation. For perceived behavioral control, the SDBT component employs a progressive difficulty structure and real-time movement guidance to lower the perceived difficulty of performing the exercises.

The program was reviewed and revised by five experts in sports rehabilitation, medical psychology, geriatrics, health management, and nursing. Additionally, a pilot study was conducted prior to the main study to assess the feasibility of the intervention. The static-dynamic balance training component was derived from balancing postural control movements, with a gradual increase in intensity by varying sensory inputs and external distractions, and consisted of three parts: (1) a 10-minute warm-up phase (including range-of-motion exercises for the wrists, hips, shoulders, knees, and ankles); (2) a 15-minute static balance training session (standing on both feet; standing in parallel and tandem; standing in tandem; standing on one foot); and (3) a 25-minutes of dynamic balance training (normal gait; narrow gait; overlapping gait; tandem gait). RT is based on Erikson's theory of psychosocial development, which states that recalling life experiences can help rural older adults resolve the psychological crisis of integration and despair in the final stages of life. Therefore, a structured procedure of reviewing the past, returning to the present, evaluating the past, and facing the present was set up and, combined with the temporal characteristics of older Chinese people's lives, recreational activities, and traditional cultural practices; reminiscence therapy involves six themes: "Our Time," "My Happy Times," "Achievements in my life," "Revisiting Traditional Festivals," "My Hobbies," and "Feeling the good old days," promoting their self-integrity and optimism to face reality with positive goal orientation. Table 1 provides the content of the SDBT-RT.

Each group of interveners consists of general practitioners, community health workers and medical postgraduate students who have undergone one month of specialized training. Thirty-two people in the intervention group were randomly divided into 8-person groups, and the appropriate time periods (8:00-10:00) were selected according to the activity habits of the elderly in the community. The intervention sites are fixed as community activity centers equipped with multimedia facilities and green rest areas. The intervention lasted for 12 weeks. In odd-numbered weeks, a dual intervention model of "40-minute RT + 50-minute SDBT" was adopted to establish behavioral intentions, and behavioral attitudes and subjective norms were strengthened through RT. Synchronous balance training enhances perceptual behavioral control through immediate improvement of physical functions. In even weeks, only 50 minutes of SDBT is conducted. A single training can reduce cognitive load and focus on the solidification of motor skills. To record engagement in reminiscence therapy, a standardized observation checklist and participant feedback forms were used after each session to assess participation and emotional responses. Facilitators were trained to recognize distress or fatigue, with activities adapted to individual conditions and emergency protocols in place for physical or psychological incidents.

The implementer is required to fill out the "Implementation Fidelity Checklist" immediately after each session, recording whether the RT theme is carried out as per the weekly plan, whether the SDBT training is upgraded in stages, and the duration of the core links. The project supervisor randomly selects 20% of the checklists every week for phone review. When deviations are found, the implementers are required to explain the reasons and formulate improvement measures at the weekly regular meeting. Meanwhile, the implementers also need to record the physical and mental states of the participants and use resources such as unified theme audio and video, handicraft materials, festival decorations and life goal lists. During the intervention period, the intervention coordinator recorded the attendance of each participant in each course and promptly followed up on those who were absent to arrange make-up classes as much as possible. A "Behavior Log Form" was designed to record changes such as supplement use, recreational activities, and disease conditions. It was reviewed monthly by general practitioners to ensure that the intervention effect was not interfered with by confounding factors. During the 4-week follow-up, participants in the intervention group received four brief weekly phone calls (5-10 minutes each) to check on home practice adherence, provide encouragement, and answer basic questions. No new intervention content was introduced.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 60 years; (2) Independent walking ability for ≥ 15 consecutive minutes (without assistive devices); (3) Long-term rural residency (≥ 1 year); (4) Provided informed consent and willingness to cooperate

Exclusion Criteria:

* (1) a diagnosis of severe pre-existing physical illnesses, defined as conditions that significantly impair physical functioning or require regular medical intervention (e.g., advanced heart disease, cancer, or other major organ diseases); (2) cognitive impairment (Short Portable Mental Status Questionnaire score ≥ 3); (3) taking psychotropic medication; (4) participating in psychosocial /sports interventions and (5) severe visual or hearing impairment, as determined by the medical records.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
The Healthy Aging Instrument (HAI) | One month
  The Healthy Aging Instrument (HAI) was developed by Thiamwong et al. and consists of 35 entries in 9 dimensions: Staying Cognitively Active, Staying Physically Active, Having Social Participation, Having Social Relationships and Support, Practicing Self-Care and Self-Awareness, Accepting Aging, Being Self-Sufficient and Living Simply, Making Merit and Good Deeds, and Managing Stress. A 5-point Likert scale was used (1 = not at all consistent, 2 = slightly consistent, 3 = not sure, 4 = moistening, physical functioning, social participation, social relationships and support, self-care, acceptance consistent, 5 = completely consistent). Total scores ranged from 35 to 175, with higher scores reflecting better levels of healthy aging, including more active engagement, stronger self-care, and greater psychosocial well-being. The Cronbach's α in the Chinese version was 0.93, and the internal consistency was good

CONTACTS AND LOCATIONS:
Locations (1):
- Huzhou university, Huzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No